CLINICAL TRIAL: NCT02648659
Title: The Pilot Study on Tailored Eradication Therapy According to Clarithromycin Resistance in Helicobacter Pylori Patients
Brief Title: The Pilot Study on Tailored Eradication Therapy According to Clarithromycin Resistance in H.Pylori Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Seong Woo Jeon, Associated Professor, Kyungpook National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KNUMC-JSW-ILA01
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer | interventions — ilaprazole; Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- triple with clarithromycin (Experimental): Ilaprazole 10mg qid, Amoxicillin 500mg qid, Clarithromycin bid for 2 weeks
  Interventions: Drug: Ilaprazole; Drug: Amoxicillin; Drug: Clarithromycin
- triple with metronidazole (Experimental): Ilaprazole 10mg qid, Amoxicillin 500mg qid, Metronidazole 500mg tid for 2 weeks
  Interventions: Drug: Ilaprazole; Drug: Amoxicillin; Drug: Metronidazole
- quadruple (Experimental): Ilaprazole 10mg qid, Amoxicillin 500mg qid, Clarithromycin 500mg bid, Metronidazole 500mg tid for 2 weeks
  Interventions: Drug: Ilaprazole; Drug: Amoxicillin; Drug: Clarithromycin; Drug: Metronidazole

INTERVENTIONS:
Drug: Ilaprazole — Ilaprazole 10mg 1tablet qid(4 times/day)
  Other Names: Noltec®
Drug: Amoxicillin — Amoxicillin 500mg 1capsule qid(4times/day)
  Other Names: Pamoxin®
Drug: Clarithromycin — Clarithromycin 500mg 1tablet bid(2times/day)
  Other Names: Clafaxin®
  Arms: quadruple; triple with clarithromycin
Drug: Metronidazole — Metronidazole 250mg 2tablets tid(3times/day)
  Other Names: Flasinyl®
  Arms: quadruple; triple with metronidazole

SUMMARY:
This study assessed the effect of tailored eradication therapy according to Clarithromycin resistance in Helicobacter pylori patients.

DETAILED DESCRIPTION:
This study assessed the effect of tailored eradication therapy according to Clarithromycin resistance in Helicobacter pylori patients.

The patients with gastric or duodenal ulcer by endoscopy were registered at the study and inspected Rapid Urease test, Biopsy, IgG-Hp antibody.

The tailored eradication therapy was prescribed to patients that confirmed Helicobacter pylori positive in two or more of among the three tests for 14 days. Through this, This study is to assess the effectiveness of eradication rate and to evaluate safety and tolerability of Ilaprazole 10mg qid treatment

ELIGIBILITY:
Inclusion Criteria:

* • 20 year old ≤ Male or female < 80 year old

  * Among Patients with gastric or duodenal ulcer by endoscopy, Subject who is identified Helicobacter pylori-positive in the conduct of two or more of the following tests ; Rapid Urease test, Biopsy test, IgG-Hp antibody test.
  * Subject who fully understands conditions of clinical trial
  * Subject who agrees to participate and spontaneously sign the ICF

Exclusion Criteria:

* Known hypersensitivity to experimental and concomitant drugs
* Subjects who are taking contraindicated medications for experimental and concomitant drug.
* Subjects with abnormal levels in the laboratory tests

  * Total Bilirubin, Creatinine> 1.5 times upper limit of normal
  * AST, ALT, Alkaline phosphatase, BUN> 2 times upper limit of normal
* Administrated of PPI, antibiotic medication within 2 weeks prior to commencement of the study.
* Pregnant and/or lactating women
* Reproductive aged women not using contraception
* Uncontrolled diabetics
* Uncontrolled hypertension
* Uncontrolled liver dysfunction
* Alcoholics
* Subjects with a history or possibility of digestive malignancy within 5 years
* Subjects with a history of gastrectomy or esophagectomy
* Subjects with hereditary diseases such as Galactose intolerance, Lapp lactose deficiency, glucose-galactose malabsorption
* Subjects participating in a clinical trial before another trial within 30 days
* Inconsistence judged subject by researcher

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2017-01-06 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
Eradication rate after tailored therapy assessed by urea breath test | Test at 4 -6 weeks after completion of medication
  After completion of 14days tailored therapy, the participants will be followed at 4-6 weeks with urea breath test (UBT). The eradication rate will be assessed by the result of UBT.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by questionnaire | Questionnaire and diary during medication for 14days
  During the medication of tailored therapy, the participants will be asked to check the compliance and adverse events with diary and questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Seong Woo Jeon, Principal Investigator — Kyungpook national university medical center

IPD SHARING:
Plan to Share IPD: No